CLINICAL TRIAL: NCT05244785
Title: Investigation on Nutritional Health and Growth Status of Primary and Middle School Students in Shenzhen, 2021
Brief Title: Health and Nutrition Survey on Shenzhen Children
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Chronic Disease Control (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Ji-Chang, Asso. Prof., Shenzhen Center for Chronic Disease Control
Other Study IDs: Child2021
Record Dates: First submitted 2021-10-28; First posted 2022-02-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Nutrition Disorder, Child; Nutrition Disorders in Adolescence; Nutritional Deficiency; Nutrition, Healthy; Nutritional Stunting; Nutritional and Metabolic Diseases; Nutritional Imbalance; Development, Child; Development, Adolescent; Growth Disorders; Growth; Stunting, Nutritional
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition; Nutritional and Metabolic Diseases; Growth Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Master and analyze the nutritional health, growth and development status of primary and secondary school students in Shenzhen, and discover the main nutritional health, growth and development problems and influencing factors.
2. Provide basic data and evidence-based basis for the municipal government and related departments to formulate child health policies and measures.

ELIGIBILITY:
Inclusion Criteria:

With signed consent to be a study subject.

Exclusion Criteria:

None.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primary and secondary school students in Shenzhen.
Sampling Method: Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Weight | 6 months
  kg
Height | 6 months
  cm
Blood pressure | 6 months
  mmHg
Vitamin concentrations in circulation | 8 months
  measured by EIA, CLIA or LC-MS/MS, nmol/L
Mineral concentrations in circulation | 8 months
  measured by ICP-MS, mass/volume
Glucose and lipid concentrations in circulation | 6 months
  measured by biochemical analyzer, mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jingfan Xiong, Director, Principal Investigator — Shenzhen Center for Chronic Disease Control
Locations (1):
- Shenzhen Center for Chronic Disease Control, Shenzhen, Guangdong, China